CLINICAL TRIAL: NCT05700227
Title: Daily Online Adaptive Short-Course Radiation Therapy and Concurrent Chemotherapy for Muscle-Invasive Bladder Cancer: A Prospective Trial of an Individualized Approach for Reducing Bowel and Bladder Toxicity (ARTIA-Bladder)
Brief Title: Daily Online Adaptive Short-Course Radiation Therapy and Concurrent Chemotherapy for Muscle-Invasive Bladder Cancer
Acronym: ARTIA-Bladder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2021-05
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Muscle Invasive Bladder Urothelial Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Daily Adaptive External Beam Radiation Therapy (Experimental): Daily adaptive radiation therapy delivered with Varian Ethos treatment system
  Interventions: Radiation: Daily Adaptive External Beam Radiation Therapy

INTERVENTIONS:
Radiation: Daily Adaptive External Beam Radiation Therapy — Daily adaptive external beam radiation therapy delivered on Varian Ethos treatment system.

SUMMARY:
This trial is a single-arm, prospective, multi-center clinical trial designed to demonstrate that adaptive radiotherapy for muscle-invasive bladder cancer will translate into a decreased rate of acute (assessed weekly during chemo-radiotherapy) grade 3 or greater gastrointestinal/genitourinary toxicity compared with the historically reported rate for non-adaptive radiation therapy. The Common Terminology Criteria for Adverse Events (CTCAE) version 5 assessment tool will be utilized.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients must have histologically proven cT2-T4aN0M0 (AJCC v8) urothelial carcinoma of the bladder with an intact bladder. Mixed urothelial histology is permitted as long as there is some urothelial histology component and no small cell component present.
3. Patients must have undergone an attempt at maximal transurethral resection of bladder tumor (TURBT) within 70 days prior to enrollment.
4. A negative pelvic nodal status is to be confirmed by one or more of the following studies/procedures: PET/CT scan, CT scan, MRI scan, fine needle biopsy, extra peritoneal biopsy, or laparoscopic biopsy, per institutional standard of care.
5. Patients must be planning to undergo concurrent pelvic radiation and chemotherapy with curative intent.
6. ECOG performance status ≤2 (Karnofsky ≥60%).
7. Ability to complete required patient questionnaires.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Patients must have normal organ and marrow function as defined below, obtained within 28 days prior to enrollment:

   * absolute neutrophil count ≥1,500/mcL
   * platelets ≥100,000/mcL
   * hemoglobin ≥9 g/dL (can be transfused with red blood cells pre-study)
   * total bilirubin ≤1.5 × institutional upper limit of normal (ULN) unless the patient has Gilbert's syndrome who must have total bilirubin <3.0 mg/dL
   * AST(SGOT)/ALT(SGPT) ≤3 × ULN
   * alkaline phosphatase ≤2.5 × ULN
   * creatinine clearance ≥30 ml/min. We recommend avoiding cisplatin for patients with creatinine clearance <50 ml/min.

   For the purpose of estimating the creatinine clearance, this formula may be used:

   Estimated creatinine clearance=((140-age)×wt (kg) ×0.85 (if female))/(72 x creatinine (mg/dl) )
10. Female patients of childbearing potential (defined as having a menses at any time in the preceding 12 months) must have a negative serum pregnancy test prior to enrollment. Patients must not be pregnant or nursing because of the potential risk of injury to the fetus/child.

Exclusion Criteria:

1. Grade ≥ 2 CTCAE GI or grade ≥ 3 GU symptoms/conditions at baseline (including ongoing refractory gross hematuria post TURBT)
2. Patients with clinically involved nodes (nodes consistent morphologically with malignancy and which are greater than 1 cm on short axis on CT or MRI).
3. Patients with cT4b disease. Patients with T4 disease after 8 subjects with T4 disease have been enrolled.
4. Bilateral hydronephrosis or diffuse carcinoma in situ based on cystoscopy or biopsy. Unilateral hydronephrosis is allowed provided the patient's kidney function meets the trial criteria. Patients should be evaluated for consideration of stenting or nephrostomy tubes for moderate-to-severe unilateral hydronephrosis prior to initiation of chemo-radiotherapy.
5. Prior radiation therapy to the pelvis or abdominal cavity, prior systemic chemotherapy/systemic therapy for bladder cancer. Prior intravesical therapy (BCG, interferon, intravesical chemotherapy) is allowed provided the time interval from completion of intravesical therapy is at least 3 months.
6. Prior cystectomy or partial cystectomy.
7. Prior malignancy (except for non-melanoma skin cancer) unless disease-free for at least 2 years. Prior non-muscle invasive bladder cancer is allowed. Patients must not have a history of urothelial carcinoma or variant histology at any site outside of the urinary bladder within the previous 24 months except Ta/T1/carcinoma in situ of the upper urinary tract (including renal pelvis and ureter) provided the patient has undergone complete nephroureterectomy and still meets trial eligibility for creatinine clearance. Patients with localized prostate cancer who are being followed on an active surveillance program are also eligible.
8. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
9. Prior systemic anticancer therapy due to a diagnosis of cancer (e.g., chemotherapy, targeted therapy, immunotherapy) within 3 years prior to entering the study or induction chemotherapy prior to the start of concurrent chemo-radiotherapy
10. Serious medical comorbidities precluding RT and/or chemotherapy (e.g., active uncontrolled infection )
11. Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease.
12. Patients with scleroderma. Patients who are symptomatic from other auto-immune diseases or patients on biologic therapies for auto-immune diseases are also excluded.
13. Patients with active tuberculosis (TB).
14. Patients who are pregnant or actively breastfeeding and who do not agree to discontinue breastfeeding before the initiation of radiation treatment planning or bladder cancer therapy.
15. Women of childbearing potential and men who do not agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of protocol treatment, and for 5 months after the last study treatment.
16. Patients with a prior known history or current diagnosis of bowel fistula.
17. Patients who undergo a pelvic or para-aortic lymph node dissection prior to planned chemoradiation therapy.
18. Patients with known active infection of HIV.
19. Patients with bilateral hip prosthetics. Select patients with unilateral hip prosthetics are eligible provided that a diagnostic CT scan permits good visualization of the entire bladder and adjacent bowel. Patients with poor visualization of the bladder/bowel on diagnostic CT scan prior to simulation should not be enrolled.
20. Patients with poorly visualized bladder and bowel on diagnostic CT [either due to body habitus or artifact (motion, artifact, etc.)] are excluded.
21. Patients who in the opinion of the investigator are not able to spend 30 minutes lying on the radiation therapy treatment couch due to significant urinary frequency/urgency or other co-morbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Acute GI/GU Toxicity | Assessed during the 4 weeks of external beam radiation therapy
  Acute gastrointestinal and genitourinary CTCAE v5 grade 3 or higher toxicity

SECONDARY OUTCOMES:
Loco-regional Tumor Control | From baseline to 24 months after completion of chemoradiotherapy
  Loco-regional bladder tumor control at 2 years. Events include histologically proven presence of muscle-invasive disease or clinical evidence of nodal disease
Patient-reported Quality of Life | From baseline to 24 months after completion of chemoradiotherapy
  Patient-reported quality of life changes during and after EBRT treatment using adaptive IMRT by the subscale EORTC QLQ-BLM30 and EPIC 26
Adverse Events | From the start of external beam radiation therapy to 24 months after completion chemoradiotherapy
  Physician reported CTCAE V5 adverse events
Global Function | From baseline to 24 months after completion of chemoradiotherapy
  Change in global function as measured with EuroQol 5 dimension 5 level (EQ-5D-5L) questionnaire. Higher scores for a given dimension indicate degraded function.
Disease-free Survival | From the start of external beam radiation therapy to 24 months after completion chemoradiotherapy
  Disease-free survival at 2 years (events include histologically proven presence of muscle-invasive disease, clinical evidence of nodal or metastatic disease, or death due to any cause)
Bladder Intact Event-free Survival | From the start of external beam radiation therapy to 24 months after completion chemoradiotherapy
  Bladder intact event-free survival at 2 years (events include histologically proven presence of muscle-invasive disease, clinical evidence of nodal or metastatic disease, radical cystectomy, or death due to any cause)
Bladder-cancer Specific Mortality | From the start of external beam radiation therapy to 24 months after completion chemoradiotherapy
  Bladder-cancer specific mortality at 2 years
Overall Survival | From the start of external beam radiation therapy to 24 months after completion chemoradiotherapy
  Overall survival at 2 years
NTCP Model | Assessed during the 4 weeks of external beam radiation therapy
  Normal tissue complication probability (NTCP) model of acute GI toxicity for hypofractionated bladder RT based on true integrated daily dose to the bowel
Adaptive Workflow Feasibility | Assessed during the 4 weeks of external beam radiation therapy
  Workflow feasibility of adaptive image guided EBRT for bladder cancer (including measuring time on table and frequency of using the adapted vs. original treatment plan for each fraction)
Dosimetric Coverage | Assessed during the 4 weeks of external beam radiation therapy
  Improvement in target coverage and/or reduction in dose to critical organs at risk compared to the non-adaptive planned dosimetry
Acute GI/GU Toxicity (>75% daily adaptive sub-cohort analysis) | Assessed during the 4 weeks of external beam radiation therapy
  Acute grade 3 or higher GI/GU CTCAE v5 toxicity rate in subjects who received 75% or more of their fractions as adaptive treatments
Acute GI/GU Toxicity (partial bladder boost sub-cohort analysis) | Assessed during the 4 weeks of external beam radiation therapy
  Acute GI/GU CTCAE v5 grade 3 or higher toxicity (assessed weekly during chemo-radiotherapy) in the cohort treated with partial bladder boost to 55 Gy

OTHER OUTCOMES:
Exploratory Translational Objective | From the start of external beam radiation therapy to 24 months after completion chemoradiotherapy
  To test the hypothesis that a biomarker driven genomic test, Decipher Bladder, performed on the TURBT specimen can be used as a prognostic/predictive biomarker for recurrence in patients treated with concurrent chemo-radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Brian Baumann, MD, Principal Investigator — Springfield Clinic
Locations (1):
- Washington University, St. Louis, St Louis, Missouri, United States